CLINICAL TRIAL: NCT00260468
Title: Structural and Functional Cerebral Findings in Late-Onset Major Depression
Brief Title: Brain Abnormalities in Late-Onset Major Depression
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Medical Research Council (Other); Bayer (Industry)
Responsible Party: Professor Poul Videbech, MD, DrMedSc, Centre for Psychiatric Research, Aarhus University Hospital, Risskov, Denamrk
Other Study IDs: 20051050
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Major Depression
Keywords: Major depression; Magnetic resonance imaging; White matter lesions; Perfusion; Diffusion; Magnetization transfer; Vascular risk factors
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Apolipoprotein
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Clinical examination program — Psychiatric/clinical interview MRI scan Blood samples Saliva samples Eye examination

SUMMARY:
The objective of this project is to examine the state of the brain in people over 50 years old suffering from late-onset depression by means of an extensive clinical assessment programme, including magnetic resonance imaging (MRI), neuropsychological testing, neurological examination, eye examination as well as blood and saliva samples. The results are to be compared with results from a control group matched for gender and age.

DETAILED DESCRIPTION:
Major depression is a frequent and serious disorder with different prognoses and complications with respect to lack of treatment response, recurrence and suicide.

MRI of the brain can provide information about changes in the brain tissue with depression, e.g. lesions of nerve connections, small thrombi or changes in the blood flow. These changes appear primarily after the age of 50 and are seen in cases of diabetes and high blood pressure. Furthermore, the connection between disruptions in the body's stress response system and depression will be explored, which is very important since studies indicate that stress and depression can affect certain brain parts permanently. This will give us a better understanding of the connection between brain changes, neuropsychology and depression prognosis, which is decisive for accurate diagnostics, effective treatment and targeted prevention of the disease in the long run.

The project is part of a larger clinical assessment programme in the Neuropsychiatric Unit under the Centre for Basic Psychiatric Research, Aarhus Psychiatric Hospital, Denmark, which gives us unique possibilities of combining research and daily clinical work. The hope is in the future to be able to offer patients in the risk group better assessment and treatment to prevent complications and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* first time major depression
* age over 50 years
* Caucasian
* admitted at a psychiatric hospital or treated at a local psychiatric clinic in Aarhus Amt

Exclusion Criteria:

* major brain damage (e.g. stroke, epilepsy, trauma)
* major alcohol or drug abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Subjects with first-episode late-onset major depression from psychiatric hospital or clinic
  2. Healthy controls
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2005-11; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raben Rosenberg, Professor, MD, DrMedSc, Study Director — Aarhus University Hospital; Videbech Poul, Professor, MD, DrMedSc, Principal Investigator — Aarhus University Hospital; Leif Østergaard, Professor, MD, DrMedSc, PhD, Study Chair — Center for Functionally Integrative Neuroscience (CFIN), Aarhus University Hospital, Denmark
Locations (1):
- Centre for Psychiatric Research, Aarhus University Hospital, Risskov, Denmark